CLINICAL TRIAL: NCT02035787
Title: Metformin With the Levonorgestrel-Releasing Intrauterine Device for the Treatment of Complex Atypical Hyperplasia (CAH) and Endometrial Cancer (EC) in Non-surgical Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Golfers Against Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1326; 12-0886 (Other: IRB)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Complex Atypical Hyperplasia; Endometrial Cancer
Keywords: metformin; endometrial cancer; Lineberger Comprehensive Cancer Center; complex atypical hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin, 850 mg. twice daily.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin added to standard non-surgical treatment with levonorgestrel-Releasing Intrauterine Device.
  Other Names: glucophage

SUMMARY:
Purpose: This is an open label, single-arm, single-center study of the addition of metformin to standard levonorgestrel-releasing intrauterine device (LR-IUD) treatment of 30 evaluable non-surgical patients with either complex atypical hyperplasia (CAH; n=15) or grade 1 endometrial adenocarcinoma (EC; n=15).

Participants:Women, over the age of 18 years, with biopsy-proven CAH/EC who are not candidates for surgical management, and therefore are planned to start standard of care treatment with the LR-IUD

Procedures (methods): subjects will be given oral metformin therapy for 12 months, or until disease progression occurs (whichever occurs first), in addition to LR-IUD treatment. Serial endometrial biopsies will be performed, as per standard of care, to assess disease status.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Primary Objective

-To compare the rate of CR at 6 months in non-surgical grade 1 EC and CAH patients receiving metformin + LR-IUD to 50%

Secondary Objectives

* to estimate the rate of CR at 6 months separately in grade 1 EC and CAH patients receiving metformin + LR-IUD
* to estimate the rate of CR at 12 months in non-surgical grade 1 EC and CAH patients receiving metformin + LR-IUD
* to document patient adherence to long-term (≥3 months) metformin administration
* To describe safety of metformin + LR-IUD treatment

Exploratory Objectives

* To explore changes in cellular proliferation as measured by the marker, Ki-67, from baseline to 6 months
* To explore association between the level of expression of the metformin transporter proteins and key targets of the metformin/mammalian target of rapamycin (mTOR) signaling pathway and CR status at 6 months
* To perform a comprehensive unbiased profiling of metabolites by analyzing the metabolic "fingerprints" of the biofluids (i.e. serum and urine) and "footprints" of the tumor tissue pre- and post- 6 months of metformin treatment
* To explore association between metabolic factors and metformin concentration levels in tumor tissue/blood/urine and CR at 6 months

This is an open label, single-arm, single-center study of the addition of metformin to standard levonorgestrel-releasing intrauterine device (LR-IUD) treatment of 30 evaluable non-surgical patients with either complex atypical hyperplasia (CAH; n=15) or grade 1 endometrial adenocarcinoma (EC; n=15). Women, over the age of 18 years, with biopsy-proven CAH/EC who are not candidates for surgical management, and therefore are planned to start standard of care treatment with the LR-IUD, will be given oral metformin therapy for 12 months, or until disease progression occurs (whichever occurs first), in addition to LR-IUD treatment. Serial endometrial biopsies will be performed, as per standard of care, to assess disease status. We hypothesize that the addition of metformin to standard LR-IUD treatment of CAH and grade 1 EC will result in a complete response (CR) rate at 6 months that is significantly higher than 50% in a population of non-surgical candidates. In addition, we plan to estimate CR rate at 6 months in CAH and EC separately, and in the group as a whole at 12 months. We will also document the rate of patient adherence to long-term metformin therapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria to participate in this study:

* Histologically confirmed CAH or grade 1 EC
* Females age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 4
* Non-surgical candidates due to:

  * Desire for fertility preserving treatment
  * Unacceptable surgical risk as defined by:

    * American Society of Anesthesiologists Physical Status (ASA) ≥ 4 and/or Perioperative Cardiac Risk > 5%(45) and/or Perioperative Respiratory Failure Risk > 5%(46)

AND

oIndependent medicine or cardiology pre-op consultation concluding 'high' surgical risk.

* Planned treatment with the LR-IUD for CAH or grade 1 EC by primary physician
* Women of childbearing potential (WOCBP) must have negative pregnancy test within 7 days of D1 of treatment
* Understand study design, risks, and benefits and have signed informed consent

Exclusion Criteria Any patient meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Evidence of renal dysfunction (Cr > 1.5mg/dL or Cr clearance < 60 mL/m2) or liver dysfunction (AST/alanine aminotransferase (ALT) > 2x upper limit of normal (ULN))
* Currently receiving progestin therapy (local, topical, or systemic)
* Myometrial invasion >50% or evidence of nodal or metastatic disease on baseline MRI (MRI only to be done for EC patients) or tumor size > 2cm on MRI or pelvic ultrasound
* Mixed histology including clear cell, serous, undifferentiated or sarcomatous elements
* Prior or current use of metformin within the past 3 months
* History of hypersensitivity to metformin or history of discontinuation secondary to attributed adverse effects
* Chronic (daily use for > 1 month) use of cimetidine (significant increase in metformin concentration and risk of lactic acidosis)
* Iodinated contrast agents used in prior 48 hours (significant increase in metformin concentration and risk of lactic acidosis)
* Pregnant or lactating
* Recent (< 4 weeks) active, documented, cervical infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02-27 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - TriHealth, Cincinnati, Ohio

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the study between 02/27/2014 and 10/12/2023, at three sites in the United States.
Pre-assignment Details: Twenty participants joined the study.
Groups:
- Complex Atypical Hyperplasia: Subjects with biopsy-proven complex atypical hyperplasia
- Grade 1 Endometrial Adenocarcinoma: Subjects with biopsy-proven Grade 1 endometrial adenocarcinoma
Period: Overall Study- 12 Months
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma
Started | 12 | 8
Completed | 4 | 6
Not Completed | 8 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Complete response | 4 | 1
Not completed — Protocol Violation | 1 | 1
Period: Overall Study -6 Months
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma
Started | 12 | 8
Completed | 7 | 7
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Population: Subjects with biopsy-proven complex atypical hyperplasia or grade 1 endometrial carcinoma.
Groups:
- Total: Total of all reporting groups
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (16.77) | 42.75 (17.87) | 41.4 (16.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate - 6 Months
Description: Complete Response is subjects with complex atypical hyperplasia or Grade 1 endometrial adenocarcinoma percentage of individuals achieved complete disease regression as defined by no evidence of microscopic viable hyperplasia or carcinoma on endometrial biopsy.
Time Frame: Up to 6 months
Population: Subjects who are with complex atypical hyperplasia or Grade 1 endometrial adenocarcinoma, started the study treatment, and an endometrial biopsy was performed to assess the treatment response, regardless of completion of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Whole Group: Subjects with complex atypical hyperplasia or Grade 1 endometrial adenocarcinoma.
Arm/Group | Whole Group
Number analyzed (Participants) | 15
percentage of participants | 80 [52 to 96]

2. Secondary Outcome: Complete Response Rate by Group
Description: Complete Response is the percentage of individuals achieving complete disease regression as defined by no evidence of microscopic viable hyperplasia or carcinoma on endometrial biopsy in complex atypical hyperplasia and Grade 1 endometrial adenocarcinoma groups. The group are based on the initial treatment assignment and not on the treatment eventually received.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma
Number analyzed (Participants) | 10 | 5
percentage of participants | 100 [72 to 100] | 40 [5 to 85]

3. Secondary Outcome: Percent Complete Response Rate-12 Months
Description: Complete Response is the percentage of participants achieving complete disease regression as defined by no evidence of microscopic viable hyperplasia or carcinoma on endometrial biopsy.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Complex Atypical Hyperplasia: Subjects with complex atypical hyperplasia.
- Grade 1 Endometrial Adenocarcinoma.: Subjects with Grade 1 endometrial adenocarcinoma.
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma.
Number analyzed (Participants) | 11 | 5
percentage of participants | 100 [74 to 100] | 60 [23 to 88]

4. Secondary Outcome: Adherence of Treatment
Description: Patients adhered to at least 80% of the scheduled doses throughout the prescribed treatment period. Subjects who achieved a biopsy-proven complete response stopped the treatment early but were still considered adherent to the treatment.
Time Frame: 12 months
Population: Subjects who are with complex atypical hyperplasia or Grade 1 endometrial adenocarcinoma, started the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma
Number analyzed (Participants) | 11 | 7
Participants | 10 | 7

5. Secondary Outcome: Treatment Attributed Adverse Events
Description: All treatment-attributed adverse events (definite, possible, and probable) with grade information are reported based on The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  CTCAE is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to 12 months
Population: Subjects who are with complex atypical hyperplasia or Grade 1 endometrial adenocarcinoma, started the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma.
Number analyzed (Participants) | 12 | 8
Participants
  Abdominal pain Grade1 | 0 | 1
  Abdominal pain Grade 2 | 0 | 1
  Alanine aminotransferase increased Grade1 | 2 | 1
  Alanine aminotransferase increased Grade 2 | 0 | 1
  Anorexia Grade1 | 2 | 1
  Anxiety Grade2 | 1 | 1
  Aspartate aminotransferase increased Grade1 | 2 | 1
  Aspartate aminotransferase increased Grade2 | 0 | 1
  Blood and lymphatic system disorders - Other, specify Grade1 | 2 | 1
  Blood and lymphatic system disorders - Other, specify Grade2 | 0 | 1
  Diarrhea Grade 1 | 4 | 3
  Diarrhea Grade 2 | 2 | 1
  Diarrhea Grade 3 | 1 | 0
  Dizziness Grade 2 | 1 | 1
  Headache Grade1 | 1 | 0
  Headache Grade2 | 1 | 0
  Fatigue Grade1 | 0 | 1
  Insomnia Grade1 | 0 | 1
  Nausea Grade1 | 8 | 4
  Nausea Grade2 | 2 | 0
  Reproductive system and breast disorders - Other, specify Grade1 | 1 | 0
  Stomach pain Grade1 | 0 | 1
  Vaginal hemorrhage Grade1 | 1 | 0
  Vaginal discharge Grade1 | 0 | 1
  Vomiting Grade 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 13 months
Description: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment. Any hospital admission was graded as a serious adverse event per protocol.
Arm/Group | Complex Atypical Hyperplasia | Grade 1 Endometrial Adenocarcinoma
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/8
Other Adverse Events (participants affected / at risk) | 12/12 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Complex Atypical Hyperplasia (N=12) | Grade 1 Endometrial Adenocarcinoma (N=8)
Renal calculi (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Complex Atypical Hyperplasia (N=12) | Grade 1 Endometrial Adenocarcinoma (N=8)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 4
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Rhinitis infective (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Creatinine increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Renal calculi (Renal and urinary disorders) | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT02035787/Prot_SAP_000.pdf